CLINICAL TRIAL: NCT03632369
Title: Hyperpolarized Noble Gas MRI Detection of Radiation-Induced Lung Injury
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled and no data was collected for the study
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Collaborators: NOAMA (Unknown)
Responsible Party: Sponsor
Other Study IDs: RP-429-01112016
Record Dates: First submitted 2018-06-21; First posted 2018-08-15 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Radiation Induced Lung Injury; Non Small Cell Lung Cancer
Keywords: MRI; Hyperpolarized; xenon-129
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Optimization Group: The primary objective of this study is to determine an optimized set of scan parameters for HP 129Xe MR diffusion-weighted imaging, HP 129Xe MR ventilation imaging, HP 129Xe Chemical Shift Saturation Recovery (CSSR) and Xenon polarization Transfer Contrast (XTC) MRI that will produce clear, anatomically and clinically relevant images of the lungs in up to 10 healthy participants and up to 10 participants with NSCLC. The primary objective will be completed before moving onto the secondary objective.
  Interventions: Diagnostic Test: Hyperpolarized xenon-129 MRI
- Delineate Functional vs. non-functional lung tissue: The secondary objective of this study is to delineate functional versus non-functional lung tissue and the effects of radiotherapy. This objective will be explored by performing these five optimized techniques with up to 10 participants with NSCLC at three time points: before radiotherapy begins, at the end of radiotherapy, and at least 10-weeks post-radiation treatment. These results will be correlated with those from PFTs and CT scans performed at corresponding time points.
  Interventions: Diagnostic Test: Hyperpolarized xenon-129 MRI

INTERVENTIONS:
Diagnostic Test: Hyperpolarized xenon-129 MRI — Participants will be asked to inhale the xenon-129 contrast agent according to procedure for gas administration. The success criterion of the drug is a obtained Xe MRI lung image with reasonable signal level. The clinical MRI scanner Philips Achieva 3.0T will be equipped with 129Xe Quadrature Transreceive Lung Coil (Large and Small) to acquire 129Xe lung images. The resonator length of the large coils is equal to 122 cm, whereas the same size of the small coil is equal to 106 cm. The success criterion of the device performance is the obtained reasonable Xe MRI lung image.

SUMMARY:
Lung cancer is the leading cause of cancer death in the world; each year lung cancer claims over 20 000 lives in Canada and more than one million lives globally (1). Significant improvements have been made in treating many other types of cancer, but lung cancer care has not realized similar successes. Seventy percent of cancers are at an advanced stage at diagnosis, and radiation plays a standard role as a part of both radical and palliative therapy in these cases. Normal lung tissue is highly sensitive to radiation. This sensitivity poses a serious problem; it can cause radiation pneumonitis or fibrosis (RILI), which may result in serious disability and sometimes death. Thirty-seven percent of thoracic cancer patients treated with radiation develop RILI; in 20% of radiation therapy cases, injury to the lungs is moderate to severe (2). In addition, radiation-induced pneumonitis that produces symptoms occurs in 5-50% of individuals given radiotherapy for lung cancer (3, 4).

The chances of clinical radiation pneumonitis are directly related to the irradiated volume of lung (5). However, radiation planning currently assumes that all parts of the lung are equally functional. Identification of the areas of the lung that are more functional would be beneficial in order to prioritize those areas for sparing during radiation planning. In order to limit the amount of RILI to preserve lung function in patients, clinicians plan radiation treatment using conformal or intensity-modulated radiotherapy (IMRT). This makes use of computed tomography (CT) scans, which take into account anatomic locations of both disease and lung but cannot assess the functionality of the lung itself. An important component of the rationale of IMRT is that if doses of radiation entering functional tissue are constrained, radiation dose can be focused on tumours to spare functional tissues from injury to preserve existing lung function (6). Therefore, to optimally reduce toxicity, IMRT would depend on data of not only tumour location, but also regional lung function.

Pulmonary function tests (PFTs) can detect a decrease in pulmonary function due to the presence of tumours or RILI, but because the measurements are performed at the mouth, PFTs do not provide regional information on lung function. Positron emission tomography (PET) imaging may be used for radiation planning, but PET is limited in its ability to delineate functional tissue, it requires administration of a radiopharmaceutical agent, it is a slow modality, and, because it requires use of a cyclotron, it is expensive. Single-photon emission computed tomography (SPECT) imaging to measure pulmonary perfusion as a means for delineating functional tissue has been explored (7-11). Whereas SPECT can detect non-functional tissue, it offers spatial resolution that is only half that of CT or PET, and it does not possess the anatomical resolution necessary for optimal use with IMRT. Furthermore, like PET, SPECT is a slow modality. Given the limitations of existing imaging modalities, there is an urgent unmet medical need for an imaging modality that can provide complimentary data on regional lung function quickly and non-invasively, and that will limit tissue toxicity in radiotherapy for non-small cell lung cancer (NSCLC).

Hyperpolarized (HP) gas magnetic resonance imaging (MRI) has the potential to fill this unmet need. HP gas MRI, uses HP xenon-129 (129Xe) to provide non-invasive, high resolution imaging without the need for ionizing radiation, paramagnetic, or iodinated chemical contrast agents. HP gas MRI offers the tremendous advantages of quickly providing high-resolution information on the lungs that is noninvasive, direct, functional, and regional. Conventional MRI typically detects the hydrogen (1H) nucleus, which presents limitations for lung imaging due to lack of water molecules in the lungs. HP gas MRI detects 129Xe nuclei, which are polarized using spin-exchange optical pumping (SEOP) technique to increase their effective MR signal intensity by approximately 100,000 times. HP gas MRI has already been widely successful for pulmonary imaging, providing high-resolution imaging information on lung structure, ventilation function, and air-exchange function. The technology has proven useful for imaging asthma, chronic obstructive pulmonary disease (COPD), and cystic fibrosis, and for assessing the efficacy of therapeutics for these diseases (12 -21). In this project, the investigators propose to develop an imaging technology for delineating regions of the lung in humans that are non-functional versus those that are viable; using hyperpolarized (HP) xenon-129 (129Xe) magnetic resonance imaging (MRI), will better inform beam-planning strategies, in an attempt to reduce RILI in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Is either:

   1. A healthy volunteer (i.e. someone not diagnosed with NSCLC; this cannot include smokers who have not been diagnosed with a lung disorder), or
   2. Has been diagnosed with NSCLC
3. Able to provide informed consent
4. Able to hold their breath for imaging

   1. Healthy volunteers enrolled in this study must be able to hold their breath for 25 seconds.
   2. Participants with NSCLC must be able to hold their breath for 15 seconds.

Exclusion Criteria:

1. Have contraindication to MR imaging (i.e. ferrous implants, cardiac pacemakers) - determined by MR screening prior to scans.
2. Have a history of claustrophobia.
3. Female exclusion only: are or may be pregnant, or are planning to become pregnant.
4. Requires an oxygen mask and cannot use a nasal cannula.
5. Blood oxygen saturation is below 92% (measured at rest in a sitting position, and with an O2 nasal cannula if the participant normally uses one).
6. Has had an acute respiratory infection in the past 10 days.
7. Is a student currently enrolled in a course at Lakehead University where the Principal Investigator (PI) is the instructor.
8. Is a student currently enrolled in a degree program at Lakehead University where the PI is their direct thesis supervisor.
9. Is currently an employee of the PI at the Thunder Bay Regional Health Research Institute (TBRHRI) and/or Lakehead University.

Healthy Volunteer Exclusion Criteria

1. Must be a non-smoker (self-identified)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve healthy participants as well as participants with NSCLC from Thunder Bay and the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Delineate functional vs. non-functional lung tissue | Before radiotherapy
  Performing HP 129Xe MR diffusion-weighted imaging, HP 129Xe MR ventilation imaging, HP 129Xe CSSR and XTC MRI the location of functional and non-functional lung tissue will be determined, and the radiotherapy will be planned based on the obtained tissue distributions. MRI results will be correlated with PFTs and CT scans.
Measure changes caused by radiotherapy in the lung tissue | At the end of radiotherapy (up to 13 months after the beginning of the study) and 10-weeks post-radio-therapy
  Performing HP 129Xe MR diffusion-weighted imaging, HP 129Xe MR ventilation imaging, HP 129Xe CSSR and XTC MRI results will be correlated with those from PFTs and CT scans performed at corresponding time points to determine the effects of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Albert, PhD, Principal Investigator — Thunder Bay Regional Health Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2015. Toronto, ON: Canadian Cancer Society; 2015. 2. Mathew L, Wheatley A, Castillo R, Castillo E, Rodrigues G, Guerrero T, Parraga G. Hyperpolarized (3)He magnetic resonance imaging: comparison with four-dimensional x- ray computed tomography imaging in lung cancer. Acad Radiol. 2012;19(12):1546-1553. 3. Marks LB, Yu X, Vujaskovic Z, Small W Jr, Folz R, Anscher MS. Radiation-induced lung injury. Semin Radiat Oncol. 2003;13(3):333-345. 4. Mehta V. Radiation pneumonitis and pulmonary fibrosis in non-small-cell lung cancer: pulmonary function, prediction, and prevention. Int J Radiat Oncol Biol Phys. 2005; 63:5-24. 5. Graham MV, Purdy JA, Emami B, Harms W, Bosch W, Lockett MA, Perez CA. Clinical dose-volume histogram analysis for pneumonitis after 3D treatment for non-small cell lung cancer (NSCLC). Int J Radiat Oncol Biol Phys 1999;45(2):323-329. 6. Govaert SL, Troost EG, Schuurbiers OC, de Geus-Oei LF, Termeer A, Span PN, Bussink J. Treatment outcome and toxicity of intensity-modulated (chemo) radiotherapy in stage III non-small cell lung cancer patients. Radiat Oncol. 2012;7(1):150. [Epub ahead of print] 7. Marks LB, Spencer DP, Bentel GC, Ray SK, Sherouse GW, Sontag MR, Coleman RE, Jaszczak RJ, Turkington TG, Tapson V, et al. The utility of SPECT lung perfusion scans in minimizing and assessing the physiologic consequences of thoracic irradiation. Int J Radiat Oncol Biol Phys. 1993;26(4):659-668. 8. Christian JA, Partridge M, Nioutsikou E, Cook G, McNair HA, Cronin B, Courbon F, Bedford JL, Brada M. The incorporation of SPECT functional lung imaging into inverse radiotherapy planning for non-small cell lung cancer. Radiother Oncol. 2005;77(3):271- 277. 9. McGuire SM, Zhou S, Marks LB, Dewhirst M, Yin FF, Das SK. A methodology for using SPECT to reduce intensity-modulated radiation therapy (IMRT) dose to functioning lung. Int J Radiat Oncol Biol Phys. 2006;66(5):1543-52. 10. Shioyama Y, Jang SY, Liu HH, et al. Preserving functional lung using perfusion imaging and intensity-modulated radiation therapy for advanced-stage non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 2007;68(5):1349-58. 11. Lavrenkov K, Christian JA, Partridge M, Niotsikou E, Cook G, Parker M, Bedford JL, Brada M. A potential to reduce pulmonary toxicity: the use of perfusion SPECT with IMRT for functional lung avoidance in radiotherapy of non-small cell lung cancer. Radiother Oncol. 2007;83(2):156-162. 12. Tzeng YS, Hoffman E, Maurer R, Mansour J, Shah N, Tschirren J, Albert M. Comparison of airway diameters measurements from an anthropomorphic airway tree phantom using hyperpolarized 3He MRI and high resolution computed tomography. Magn Reson Med. 2007;58:636-642. 13. Tzeng YS, Hoffman E, Cook-Granroth J, Gereige J, Mansour J, Washko G, Cho M, Stepp E, Lutchen K, Albert M. Investigation of hyperpolarized 3He magnetic resonance imaging utility in examining human airway diameter behavior in asthma through comparison with high-resolution computed tomography. Acad Radiol. 2008;15:799-808. 14. Tzeng Y-S, Gereige J, Mansour J, Shah N, Zhou X, Washko G, Stepp E, Cho M, Szender JB, Sani SZ, Israel E, Lutchen K, Albert M. The difference in ventilation distribution and ventilation heterogeneity between asthmatic and healthy subjects quantified from hyperpolarized 3He MRI. J Appl Physiol. 2009a;106(3):813-822. 15. Tzeng YS, Lutchen K, Albert M. The difference in ventilation heterogeneity between asthmatic and healthy subjects quantified using hyperpolarized 3He MRI. J Appl Physiol. 2009b;106:813- 822. 16. Campana L, Kenyon J, Zhalehdoust-Sani S, Tzeng YS, Sun Y, Albert M, Lutchen KR. Probing airway conditions governing ventilation defects in asthma via hyperpolarized MRI image functional modeling. J Appl Physiol. 2009;106:1293-300. 17. Lee EY, Sun Y, Zurakowski D, Hatabu H, Khatwa U, Albert MS. Hyperpolarized 3He MR imaging of the lung: normal range of ventilation defects and PFT correlation in young adults. J Thorac Imaging. 2009;24:110-114. 18. Kirby M, Mathew L, Wheatley A, Santyr GE, McCormack DG, Parraga G. Chronic obstructive pulmonary disease: longitudinal hyperpolarized (3)He MR imaging. Radiology. 2010a;256(1):280-289. 19. Mullally W, Betke M, Albert M, Lutchen K. Explaining clustered ventilation defects via a minimal number of airway closure locations. Ann Biomed Eng. 2009;37:286-300. 20. Sun Y, Butler JP, Lindholm P, Walvick RP, Loring SH, Gereige J, Ferrigno M, Albert MS. Marked pericardial inhomogeneity of specific ventilation at total lung capacity and beyond. Respir Physiol Neurobiol. 2009;169:44-49. 21. Sun Y, O'Sullivan BP, Roche JP, Walvick R, Reno A., Shi L., Baker D., Mansour JK, Albert MS. Using hyperpolarized 3He MRI to evaluate treatment efficacy in cystic fibrosis patients. J Magn Reson Imaging. 2011;34(5):1206-1211.